CLINICAL TRIAL: NCT07036601
Title: A Multicenter, Randomized, Double-blind, Placebo-Parallel Controlled, Phase II Study to Evaluate the Efficacy and Safety of THDBH120 Injection in Overweight or Obese Subjects
Brief Title: Phase II Study of THDBH120 Injection in Overweight or Obese Subjects
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THDBH120L202
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Overweight or Obese
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THDBH120 injection (Experimental)
  Interventions: Drug: THDBH120 injection
- Placebo of THDBH120 injection (Placebo Comparator)
  Interventions: Drug: Placebo of THDBH120 injection

INTERVENTIONS:
Drug: THDBH120 injection — Participants received THDBH120 by subcutaneous injection.
  Arms: THDBH120 injection
Drug: Placebo of THDBH120 injection — Participants received placebo by subcutaneous injection.
  Arms: Placebo of THDBH120 injection

SUMMARY:
To assess the efficacy and safety of THDBH120 injection compared with placebo in weight reduction in overweight or obese subjects after 26 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 to 75 years of age, inclusive;
* Have a BMI ≥ 28 kg/m² or 24 ≤BMI< 28.0 kg/m² with at least 1 weight-related comorbidity at screening: prediabetes, hypertension, metabolic-associated fatty liver disease, dyslipidemia, weight-bearing joint pain, or obstructive sleep apnea syndrome;
* Diet and exercise control for at least 3 months before screening visit, and less than 5% self-reported change within the last 3 months.

Exclusion Criteria:

* History of diabetes;
* History of obesity attributable to endocrine diseases, monogenic mutations, or drug-induced causes, such as hypothalamic obesity, pituitary obesity, hypothyroid obesity, Cushing's syndrome, insulinoma, acromegaly, or hypogonadism; or weight gain resulting from increased non-fat mass (e.g., edema);
* Presence of uncontrolled hypertension at screening: systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg;
* A 12-lead electrocardiogram (ECG) shows any of the following at screening: heart rate <50 bpm or >100 bpm; QTcF prolongation (QT interval corrected by Fridericia's formula: QTc = QT/RR^0.33; >450 ms for males, >470 ms for females); PR interval >200 ms; presence of long QT syndrome; second- or third-degree atrioventricular block; left bundle branch block; complete right bundle branch block; Wolff-Parkinson-White syndrome; or any other condition that, in the opinion of the investigator, makes the subject unsuitable for participation in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight | Baseline, Week26

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve ≥5% Body Weight Reduction | Baseline, Week26
Percentage of Participants Who Achieve ≥10% Body Weight Reduction | Baseline, Week26
Percentage of Participants Who Achieve ≥15% Body Weight Reduction | Baseline, Week26
Percentage of Participants Who Achieve ≥20% Body Weight Reduction | Baseline, Week26
Change from baseline in waist circumference after the treatment | Baseline, Week 26
Change from baseline in BMI after the treatment | Baseline, Week 26
Change from baseline in blood pressure after the treatment | Baseline, Week 26
Change from baseline in HbA1c after the treatment | Baseline, Week 26
Change from baseline in total cholesterol after the treatment | Baseline, Week 26
Number of Participants with One or More Adverse Event(s) and Serious Adverse Event(s) | Week 30

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, China

IPD SHARING:
Plan to Share IPD: No